CLINICAL TRIAL: NCT02086201
Title: Stepped, Reward-exposure Based Therapy vs. PST in Late Life Depression
Brief Title: Comparing Engage to PST for Late Life Depression
Acronym: Engage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Pat Arean, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001739
Record Dates: First submitted 2014-02-25; First posted 2014-03-13 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Major Depression
Keywords: major depression; depression; depressive disorder; mental health; mental disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Psychological Well-Being; Mental Disorders | interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problem Solving Therapy (Active Comparator): Problem solving therapy is an evidence based psychotherapy for depression, with 30 years of research supporting its efficacy. PST focuses on the patients themselves and helps them develop skills in identifying, prioritizing, and solving problems, and thereby creates a sense of empowerment.
  Interventions: Behavioral: Problem Solving Therapy
- Engage (Experimental): Engage utilizes reward exposure consisting of the reintroduction of activities that patients once found rewarding and enjoyed, but have abandoned after they developed depression. Engage uses basic problem solving through which patients learn how to form "action plans" for pursuing rewarding activities of their choice.
  Interventions: Behavioral: Engage

INTERVENTIONS:
Behavioral: Problem Solving Therapy — PST is a behavioral intervention for depression that is delivered by trained therapists over a 9 week period. It consists of a process to help patients understand and then solve the problems in their lives they feel is contributing to their depression.
  Arms: Problem Solving Therapy
Behavioral: Engage — Engage is a weekly behavioral intervention that is delivered over a 9 week period of time by trained therapists. The focus of Engage is to help patient reconnect with activities that they have lost interest in pursuing due to depression.
  Arms: Engage

SUMMARY:
This is a non-inferiority trial of Engage, a new intervention for late-life depression, and problem solving therapy (PST). Patient participants will be randomized to either Engage or PST and receive 9 weeks of either intervention. Interview assessments will be collected at baseline and weeks 2, 4, 6, 8, 9, 26, and 36. Clinician participants, social workers from mental health agencies, will be randomized to receive training and certification in either Engage or PST.

DETAILED DESCRIPTION:
Policy reports document that evidence-based psychotherapies are rarely employed and sustained in the community. Several causes of this science to service gap have been identified. One cause, specific to behavioral interventions, is the complexity of interventions and the competencies community clinicians must acquire and sustain over time in order to deliver them. A realistic solution is to streamline behavioral interventions and tailor them to the settings and therapist skill level available in the community. In response to this need, we have developed Engage, which: 1) is streamlined on the basis of concepts and findings on the neurobiology of depression; 2) consists of psychotherapeutic and ecosystem management components of known efficacy; 3) has distilled and simplified these components so as they can be accessible to most depressed older patients and taught to larger numbers of clinicians than available therapies, e.g., Problem Solving Therapy (PST); and 4) is personalized through a structured stepped approach focusing on "reward exposure". Problem Solving Therapy is an evidenced-based intervention shown to be effective in treating late-life depression.

Three hundred (150 per site) patient participants will be randomly assigned to receive 9 sessions of either Engage or PST. Forty-two clinician participants will be randomly assigned to receive training and certification in either Engage or PST. Once certified, clinicians will be assigned a patient participant and administer their assigned intervention.

ELIGIBILITY:
Inclusion Criteria (Patient participants):

* Age ≥ 60 years
* unipolar, non-psychotic major depression (by SCID, DSM-IV)
* MADRS ≥ 20
* MMSE ≥ 24
* off antidepressants or have been on a stable dose of an antidepressant for 12 weeks and do not intend to change the dose in the next 10 weeks
* English speaking
* capacity to provide written consent

Exclusion Criteria (Patient participants):

* Presence of psychiatric diagnoses other than unipolar, non-psychotic major depression or generalized anxiety disorder
* Newly started use of psychotropic drugs (<12wks) or cholinesterase inhibitors other than mild doses of benzodiazepines
* Current active suicidal intent/plan
* Current substance abuse

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2014-05; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Depression | Measured at pretreatment and weeks 2,4,6,8,9,26 and 36
  Depression will be assessed using the Hamilton Depression Rating Scale, a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, PhD, Principal Investigator — UW; George Alexopoulos, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Medical College of Cornell University, White Plains, New York
  - University of Washington Department of Psychiatry and Behavioral Sciences, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We intend to share de-identified data once study is complete